CLINICAL TRIAL: NCT03674879
Title: Impact of Mobile Text Messaging on Follow Up Rates After Discharge From the Pediatric Emergency Department
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left facility
Sponsor: New York City Health and Hospitals Corporation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NYCHHC
Record Dates: First submitted 2016-07-19; First posted 2018-09-18 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Duty to Recontact
Keywords: Follow Up; Text Messaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phone Call (No Intervention): Follow up contact is attempted via phone call.
- Text Message (Experimental): Follow up contact is attempted via text message.
  Interventions: Other: Text Message

INTERVENTIONS:
Other: Text Message — Patient contact attempted with text message.
  Arms: Text Message

SUMMARY:
To compare the effectiveness of text message versus voice call as a method of contact for providing results of diagnostic tests and assuring ongoing care from the pediatric emergency department.

DETAILED DESCRIPTION:
The investigators plan to conduct a prospective randomized controlled trial to compare two means of contacting patients and their caregivers after discharge from the emergency department in order to provide results of tests: text messaging (intervention group) vs. telephone call (standard group).

ELIGIBILITY:
Inclusion Criteria:

* patients under the age of 18 who have had diagnostic testing without finalized results prior to discharge from the emergency department

Exclusion Criteria:

* Admitted patients
* Patients transferred to another facility
* Patients with critical values as results
* Do not have devices that can receive phone and text messages
* Cannot read English or Spanish

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2016-09; Primary Completion 2017-08 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Number of phone call or text message attempts to successful contact with study participant | Within 2 weeks.
  A study practitioner will make one attempt per business day to contact the patient or caregiver to provide test results and arrange follow-up care; the method will be determined by the study arm to which the participant is assigned. Participants in the standard practice control arm will receive a telephone call. If a call is not answered, a voice message will be left instructing the patient/parent to call the Pediatric Follow-Up Office. Participants in the intervention arm will receive a text message using the same script. A successful contact will be recorded when a practitioner speaks directly to the patient or parent/guardian via phone.

CONTACTS AND LOCATIONS:
Overall Officials: Czer Anthoney E Lim, MD, Principal Investigator — Jacobi Medical Center/Albert Einstein College of Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dudas RA, Pumilia JN, Crocetti M. Pediatric caregiver attitudes and technologic readiness toward electronic follow-up communication in an urban community emergency department. Telemed J E Health. 2013 Jun;19(6):493-6. doi: 10.1089/tmj.2012.0166. Epub 2013 Apr 9. PMID 23570276
- [Background] Horne A, Ros SP. Telephone follow-up of patients discharged from the emergency department: how reliable? Pediatr Emerg Care. 1995 Jun;11(3):173-5. doi: 10.1097/00006565-199506000-00008. PMID 7651874
- [Background] Levitt MA, Johnson S, Engelstad L, Montana R, Stewart S. Clinical management of chlamydia and gonorrhea infection in a county teaching emergency department--concerns in overtreatment, undertreatment, and follow-up treatment success. J Emerg Med. 2003 Jul;25(1):7-11. doi: 10.1016/s0736-4679(03)00131-8. PMID 12865101
- [Background] Neuner B, Fleming M, Born R, Weiss-Gerlach E, Neumann T, Rettig J, Lau A, Schoenfeld H, Kallischnigg G, Spies C. Predictors of loss to follow-up in young patients with minor trauma after screening and written intervention for alcohol in an urban emergency department. J Stud Alcohol Drugs. 2007 Jan;68(1):133-40. doi: 10.15288/jsad.2007.68.133. PMID 17149527
- [Background] Reed JL, Huppert JS, Taylor RG, Gillespie GL, Byczkowski TL, Kahn JA, Alessandrini EA. Improving sexually transmitted infection results notification via mobile phone technology. J Adolesc Health. 2014 Nov;55(5):690-7. doi: 10.1016/j.jadohealth.2014.05.004. Epub 2014 Jun 21. PMID 24962503
- [Background] Reed JL, Simendinger L, Griffeth S, Kim HG, Huppert JS. Point-of-care testing for sexually transmitted infections increases awareness and short-term abstinence in adolescent women. J Adolesc Health. 2010 Mar;46(3):270-7. doi: 10.1016/j.jadohealth.2009.08.003. Epub 2009 Oct 12. PMID 20159505